CLINICAL TRIAL: NCT00441493
Title: A Dose Finding Study of Fluvastatin for in Vivo Demonstration of Inhibiting Hepatitis C Replication in Patients Infected With Chronic Hepatitis C With Special Attention to the African-American Population.
Brief Title: Fluvastatin Versus Hepatitis C Virus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bader, Ted, M.D. (Individual)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13035; 13134
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2006-09

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; fluvastatin
MeSH Terms: conditions — Hepatitis C | interventions — Fluvastatin

INTERVENTIONS:
Drug: fluvastatin

SUMMARY:
This is a dose finding and efficacy trial for fluvastatin versus hepatitis C.

DETAILED DESCRIPTION:
Four different oral doses of fluvastatin will be used for 14 days and the viral load of hepatitis C will be measured weekly. This has been extended to different doses for 9-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HCV RNA positive

Exclusion Criteria:

* Testing positive for alcohol or marijuana

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Viral Load Reduction, Liver test changes

CONTACTS AND LOCATIONS:
Overall Officials: Ted Bader, MD, Principal Investigator — VA Medical Center and University of Oklahoma
Locations (1):
- VA Medical Center, Oklahoma City, Oklahoma, United States